CLINICAL TRIAL: NCT03503175
Title: A Novel Urinary Access System for Universal Transcatheter Cystoscopy at The Time of Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, charbel salamon, Principal Investigator; Director, Urogynecology, Atlantic Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1178748
Record Dates: First submitted 2018-04-02; First posted 2018-04-19 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Novel urinary access system (Experimental): Participants randomized to this arm will receive the novel urinary access system (CystoSureTM).
  Interventions: Device: Novel urinary access system (CystoSureTM)
- Standard Foley catheter (Active Comparator): Participants randomized to this arm will receive a standard Foley catheter and rigid cystoscopy.
  Interventions: Device: Standard Foley catheter

INTERVENTIONS:
Device: Novel urinary access system (CystoSureTM) — CystoSureTM is a silicone device that was developed by surgeons to enable easy and standardized cystoscopy. The design of the CystoSureTM catheter has separate channels for draining the bladder and performing cystoscopy, so doctors can perform a cystoscopy without removing the catheter (which can, as described above, potentially lead to a UTI).
  Arms: Novel urinary access system
Device: Standard Foley catheter — Participants randomized to this arm will receive a standard Foley catheter and standard rigid cystoscopy.
  Arms: Standard Foley catheter

SUMMARY:
Cystoscopy is a commonly performed procedure after gynecologic surgery, however, its use may increase patients' risk for acquiring urinary tract infections due to urinary tract instrumentation entry and reentry of the lower urinary tract with the cystoscope and foley catheter. Use of a novel multi-channel transurethral bladder catheter that allows for cystoscopy through a specialized port will permit cystoscopy to be performed without catheter removal. This may allow for intraoperative detection of urinary tract injuries with a reduction in both urethral manipulation and hospital-associated urinary tract infections. Other potential benefits may include a shorter procedure time and ease of use for providers.

DETAILED DESCRIPTION:
A cystoscopy is a procedure that inserts a thin tube with a light and camera through the urethra, so that the inside of the bladder can be checked for injuries. Current guidelines recommend that this is done after a hysterectomy. Normally, doing a cystoscopy requires that a patient's foley catheter (a tube inserted through the urethra and into the bladder to drain urine) gets removed and then replaced. This can potentially lead to a urinary tract infection (UTI).

CystoSureTM is a silicone device that was developed by surgeons to enable easy and standardized cystoscopy. The design of the CystoSureTM catheter has separate channels for draining the bladder and performing cystoscopy, so doctors can perform a cystoscopy without removing the catheter (which can, as described above, potentially lead to a UTI). In this study, investigators want to examine whether using a CystoSureTM catheter instead of a standard foley catheter could therefore lead to a reduced number of UTIs in hysterectomy patients. CystoSureTM is cleared by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-90
* Undergoing hysterectomy with or without concomitant procedures

Exclusion Criteria:

* Known history of urinary tract anomaly (i.e. urethral diverticulum, ureteral duplication, ectopic ureter)
* ≥3 UTIs in past 6 months
* Immunosuppressed patients
* Premeditated urologic procedure during hysterectomy surgery

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2018-07-26 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Urinary tract infections | Up to 4 weeks after surgery
  Rate of urinary tract infections (within 4 weeks of surgery) in patients undergoing cystoscopy with the novel urinary access system (CystoSureTM) versus rigid cystoscopy at the time of hysterectomy.

SECONDARY OUTCOMES:
Detection of urinary tract injuries | At the time of surgery
  Identification of urinary tract injuries due to index procedure at time of cystoscopy
Device feasibility | At the time of surgery
  Number of patients who were randomized to the novel urinary access system (CystosureTM) who could not receive the device due to technical issues (unable to insert catheter; device malfunction; surgeon preference)
Surgeon satisfaction | After the first and last patient enrolled by each surgeon, through study completion (which is estimated to be up to 24 months after enrollment begins).
  Survey will be collected from surgeons after the first and last use of CystoSureTM.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantic Urogynecology Associates, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No